CLINICAL TRIAL: NCT02875288
Title: Prospective Randomized Trial of Liposomal Versus Plain Bupivacaine in Minimally Invasive General Surgery Procedures
Brief Title: Trial of Liposomal Versus Plain Bupivacaine in Minimally Invasive General Surgery Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMCSD.2015.0067
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liposomal Bupivicaine arm (Experimental): Post procedure, infiltrate wounds with liposomal bupivacaine
  1. Liposomal Bupivacaine (Brand name Exparel) 266 milligram (mg)/20 mL to be diluted to 30 mL with normal saline
  2. 10 mL of study drug to be injected at each 10-12 millimeter (mm) trocar site and 5 mL of study drug to be injected at the 5 mm trocar sites. Typically there are two 10 mm trocar sites and three 5 mm trocar sites.
  Interventions: Drug: liposomal bupivicaine
- Plain Bupivicaine (Active Comparator): 1. Post procedure, infiltrate wounds with plain bupivicaine
  2. Plain Bupivacaine 0.25%, volume of 30 mL
  3. 10 mL of study drug to be injected at each 10-12 millimeter (mm) trocar site and 5 mL of study drug to be injected at the 5 mm trocar sites. Typically there are two 10 mm trocar sites and three 5 mm trocar sites.
  Interventions: Drug: liposomal bupivicaine

INTERVENTIONS:
Drug: liposomal bupivicaine — 1. The intervention that is being tested and who will perform the procedures; Two general surgeons will perform the procedure with either liposomal or plain bupivacaine.
  2. The treatment procedures or regimens; The treatment procedure is direct, surgical site infiltration with either liposomal or plain bupivacaine.
  3. Dosage level and justification; Liposomal Bupivacaine: 266 mg/20 mL liposomal bupivacaine diluted to 30 mL Plain Bupivacaine: 30 mL of 0.5% plain bupivacaine
  4. Route of drug administration; Surgical site infiltration
  Other Names: Exparel

SUMMARY:
Aim: To compare the postoperative outcomes after surgical infiltration with plain bupivacaine compared to liposomal bupivacaine in patients undergoing elective, minimally invasive, general surgery procedures. To the investigators knowledge, there are no head-to-head, prospective, randomized, controlled trials of plain bupivacaine versus liposomal bupivacaine to evaluate postoperative pain and return of function.

DETAILED DESCRIPTION:
The investigators current standard has been to use liposomal bupivacaine routinely for surgical infiltration which was a change from the historical practice of infiltration with lidocaine/bupivacaine, plain bupivacaine or no local anesthetic at all. The change was made due to the perceived benefits in analgesia past the 12-24 hours that plain bupivacaine was effective. It is not clear, however, that there are statistically significant benefits in terms of reduced narcotic use and length of hospital stay and improved pain control and return of function post-operatively.

Primary outcomes: The investigators will then measure narcotic use post-operatively as calculated by combining measures of patient-controlled analgesia (PCA) use for first 24 hours added to in-patient oral narcotic use (by referencing the electronic medical record (EMR)) as well as out-patient oral narcotic use as reported by patients. Subjective pain levels and pain interference scale and physical functioning scale will be evaluated pre-operatively and post-operatively with use of the Pain Assessment Screening Tool and Outcomes Registry (PASTOR) developed by the Defense and Veterans Center for Integrative Pain Management (DVCIPM) as a measure of perioperative pain and function.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or older
* American Society of Anesthesiologists (ASA) status 1, 2 or 3
* Having an elective, minimally invasive, general surgery procedure at Naval Medical Center San Diego (NMCSD)

Exclusion Criteria:

* Age: Younger than 18 years old
* Pregnant women - safety of liposomal bupivacaine has not been studied in pregnant women
* ASA status greater than or equal to 4
* Conversion to open procedure/laparotomy
* History of reaction to local anesthetics
* History of hepatic disease - local anesthetics are metabolized in the liver
* History of pre-operative/concurrent condition requiring narcotic use
* Patient not able to adhere to post-operative pain control regimen outlined in methods section

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Total post operative narcotic use in morphine equivalents. | Up to fourteen days.
  To be measured by combining measures of Patient-Controlled Analgesia pump use for the first 24 hours added to in-patient oral narcotic use (by referencing the electronic medical record (EMR) and out-patient oral narcotic use as reported by patients.

SECONDARY OUTCOMES:
Length of hospital stay post operative procedure. | up to fourteen days.
  Participants post operative procedure length of stay will be determined from the electronic medical record.
Pain level pre and post operative procedure. | Up to fourteen days.
  Baseline pain level will be gathered pre operative procedure and post operative procedure day one, seven, and fourteen through the 0 to 10 pain scale with 0 being "No Pain", 5 being "Moderate Pain", and 10 being "Worse Possible Pain".
Post operative procedure physical functioning level. | Up to fourteen days.
  Data is gathered on POP day one, seven and fourteen through the Physical Functioning Scale (PFS), which is scored from 0 to 100 with a higher scores indicating better physical function.
Number of post operative procedure adverse events. | Up to fourteen days.
  Data is gathered from the patient electronic medical record (EMR).

CONTACTS AND LOCATIONS:
Overall Officials: David P Gallus, MD, Principal Investigator — United States Naval Medical Center, San Diego
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No